CLINICAL TRIAL: NCT06484660
Title: Efficacy Of Minimally Invasive Approach In The Mucosal Advancement Flap Technique For The Surgical Treatment Of Previously Untreated Complex Perianal Fistula
Brief Title: Efficacy Of Minimally Invasive Approach In The Surgical Treatment Of Complex Perianal Fistula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Ignacio Fernandez Hurtado, Specialist in General Surgery. Specialist in Digestive Surgery, Hospital Son Llatzer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB4521/21
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Fistula Perianal
Keywords: Perianal Fistula; Mucosal Advancement Flap; Minimally Invasive Approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally Invasive Approach In The Mucosal Advancement Flap Technique (Experimental)
  Interventions: Procedure: Minimally Invasive Approach In The Mucosal Advancement Flap Technique

INTERVENTIONS:
Procedure: Minimally Invasive Approach In The Mucosal Advancement Flap Technique — Surgical treatment of complex perianal fistula. Less tissue damage. Electrocoagulation source with 75% lower power. Better de-epithelialization of the intra-sphinteric tract. More precise closure of orifice. More consistent mucosal flap

SUMMARY:
The goal of this clinical trial is to study whether the minimally invasive approach in the mucosal advancement flap technique for the treatment of complex perianal fistula improves the healing rate compared to non-minimally invasive surgery.

The main question it aims to answer is:

- Does the healing rate of patients undergoing minimally invasive approach in the mucosal advancement flap technique improve compared to patients undergoing non-minimally invasive surgery?

Researchers will also compare minimally invasive approach in the mucosal advancement flap technique to the non-minimally invasive approach in terms of postoperative pain, fecal incontinence and healing time.

Quality of life and global morbidity will also be analyzed.

Participants will:

* Undergo surgical treatment of complex perianal fistula performed by mucosal advancement flap performed by a minimally invasive technique.
* Attend control visits and fill in symptom forms one week, one month, three months and six months after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18.
* Present with a complex perianal fistula not surgically treated with curative intention.
* Present only one main fistulous tract.
* Mucosal advancement flap as the chosen technique for the treatment of the fistula.
* Patient has given informed consent to participate in the study.

Exclusion Criteria:

* Non-cryptoglandular internal fistulous orifice (IFO).
* Extrasphincteric fistula.
* Coexistence of anal fissure.
* Coexistence of hemorrhoids tributary to surgery.
* Coexistence of anal or rectal prolapse.
* Coexistence of inflammatory bowel disease.
* Coexistence of anal or colorrectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Healing rate | six months
  Healing will be measured if 4 criteria are present: no supuration or pain for more than a week, no open external fistulous orifice, no palpable trajectory, no internal fistulous orifice and no tract or collections in 3D endoanal ultrasound.

SECONDARY OUTCOMES:
Postoperative pain | one week
  Pain measured in visual analogic scale (VAS). Scale: 0 to 10. Higher scores mean a worse outcome.
Global morbidity | one month
  Clavien Dindo Scale. Scale: 1 to 5. Higher scores mean worse complications.
Quality of life score | six months
  SF 36 questionnaire. 36 items. Higher scores mean a better quality of life.
Fecal incontinence | six months
  Measured in Wexner scale. Score 0 to 20. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Son Llatzer, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No